CLINICAL TRIAL: NCT05871281
Title: Effects of Pelvic Floor Muscle Training and Electrostimulation on Women's Quality of Life and Pelvic Floor Muscle Function in Stress Urinary Incontinence
Brief Title: Electrostimulation and PFMT for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LithuanianSportsU 14
Record Dates: First submitted 2023-04-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Urinary Incontinence, Stress
Keywords: stress incontinence; pelvic floor; electrostimulation; muscle training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: This study is a four week, single blinded randomized controlled trial with pre-post design comparing PFM training group with PFM electrostimulation
Who Masked: Outcomes Assessor
Masking Description: outcomes were measured by gynecologists, intervention done by physiotherapist, who did not know measurements' results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle training group (Active Comparator): All subjects attended individual physiotherapy procedures, the duration of one of which was 60 minutes. One woman was assigned a total of 8 contact procedures over four weeks. During the individual procedures, exercises were selected and modified according to the women's ability to perform them. All women were taught correct abdominal breathing while lying down, to activate the abdominal muscles. Also, all were trained to perform Kegel exercises, explaining their benefits. In order to diversify and modify the exercises, they were performed with auxiliary means, i.e. using balls, gymnastic sticks, a bench, elastic bands, a physiotherapy wall, yoga blocks, rollers, weights and an aerial yoga band.
  Interventions: Procedure: Pelvic floor muscle exercises
- Pelvic floor muscle electrostimulation group (Experimental): Electrostimulation was performed with a Kegel 8 home elektrostymulator. The subjects were prescribed two electrostimulation programs: PO3 in the morning and PO10 in the evening. The duration of the PO3 program was 45 minutes, and was intended for general strengthening of the pelvic floor muscles. The duration of the PO10 program is 40 minutes. and it is prescribed for stress incontinence. Duration of interventions 4 week.
  Interventions: Procedure: Pelvic floor muscle exercises

INTERVENTIONS:
Procedure: Pelvic floor muscle exercises — Pelvic floor muscle exercises were performed from different body positions. Duration of interventions - 4 weeks. Frequency - 2 times per week, number of individual contact sessions - 8 .

SUMMARY:
The goal of this randomized controlled trial is to evaluate and compare the effects of electrostimulation in addition to pelvic floor muscle training and pelvic floor muscle training alone on pelvic floor muscle (PFM) function, urinary incontinence and quality of life in women with stress urinary incontinence. The main questions are:

What is the effect of electrostimulation combined with pelvic floor muscle training on pelvic floor muscle function, symptoms of urinary incontinence and quality of life in women with stress urinary incontinence? What is the effect of pelvic floor muscle training program on pelvic floor muscle function, symptoms of urinary incontinence and quality of life in women with stress urinary incontinence? Which intervention is more effective - electrostimulation with pelvic floor muscle training or pelvic floor muscle training alone?

Participants will be evaluated before and after the interventions with the following methods:

International Incontinence Counseling Questionnaire - Short Form (ICIQ-SF) Pelvic floor muscle strength and endurance will be assessed with a "Pelvexiser" perineometer.

DETAILED DESCRIPTION:
The study involved 24 women 20-49 years old who have complained of stress urinary incontinence for at least 4 weeks, who gave at least one birth vaginally and signed the consent form. Subjects were excluded if they were pregnant, were diagnosed with vaginismus, urinary tract infections, cancer, epilepsy, pelvic organ prolapse greater than stage I, skin diseases, had undergone previous pelvic floor surgeries, had heart stimulator, or metal implant and were unable to contract the PFM. Study participants were randomly divided into two groups: the I group (n=12), in which participants underwent pelvic floor muscle training (PFMT) and the II group (n=12) in which subjects received pelvic floor muscle exercises combined with electrostimulation (PFMES).Participants were evaluated before the interventions and repeated after 4 weeks. Before and after the interventions, women's quality of life (QoL) was assessed according to the International Incontinence Counseling Questionnaire - Short Form. Perineometry with Pelvexiser perineometer was used to measure pelvic floor muscle strength and endurance and vaginal resting pressure. Statistical analysis was performed by IBM SPSS Statistics 26.0 and Microsoft Excel software 365.

ELIGIBILITY:
Inclusion Criteria:

* Have given birth at least once
* Voluntary consent to participate in the study
* Do not have concomitant diseases
* Do not use hormonal drugs.

Exclusion Criteria:

* Less than three months have passed after childbirth
* Have heart implants or other metal implants
* Pregnancy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women after delivery
Enrollment: 24 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Quality of life by International Incontinence Counseling Questionnaire - Short Form (ICIQ - SF) | Change from Baseline Quality of Life at 4 weeks
  The questionnaire consists of four items and the overall score ranges from 0 to 21, with greater values indicating increased symptom severity: 0 - no symptoms of UI, 1-5 scores - mild symptoms of UI, 6-12 scores - moderate symptoms of UI, 13-18 scores - severe symptoms of UI, 19 - 21 scores - and very severe symptoms of UI.
Pelvic floor muscle strength and endurance | Change from Baseline Pelvic floor Muscle Strength and Endurance at 4 weeks
  Perineometry with Pelvexiser perineometer (mm Hg). The higher the results- the better function of pelvic floor muscle strength and endurance.
Resting vaginal pressure | Change from Baseline Resting Vaginal Prressure at 4 weeks
  Perineometry with Pelvexiser perineometer (mm Hg).

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Dudoniene, PhD, Study Chair — Lithuanian Sports University, Lithuania
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
IPD can not be shared according to signed by participants consent form.